CLINICAL TRIAL: NCT04964765
Title: Non-invasive Evaluation of New-onset Atrial Fibrillation After Cardiac Surgery The Basel CardioInsightTM - 3D Mapping (BigMap) Study
Brief Title: The Basel CardioInsightTM - 3D Mapping Study
Acronym: BigMap
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Basel, Switzerland (Other)
Collaborators: Medtronic (Industry); Freiwillige Akademische Gesellschaft (FAG) Basel (Unknown)
Responsible Party: Sponsor
Other Study IDs: 2021-01353; qu20Siegemund4
Record Dates: First submitted 2021-07-06; First posted 2021-07-16 (Actual); Last update posted 2025-04-09 (Actual); Status verified 2025-04

CONDITIONS: New-onset Atrial Fibrillation (NOAF)
Keywords: atrial fibrillation (AF); cardiac surgery; reentrant circuits; rotors; left atrial foci; pulmonary vein isolation; CardioInsightTM (CIT) - 3D Mapping technology; NOAF-maintaining foci
MeSH Terms: conditions — Atrial Fibrillation | interventions — Tomography, X-Ray Computed

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Mapping — CardioInsightTM Cardiac Mapping System is a non-invasive single beat cardiac mapping system that provides three-dimensional electroanatomic maps of the heart. The CIT vest is attached to the patient's torso for non-invasive mapping. To ensure correct and rapid mapping of the NOAF by the CIT device, it is essential to briefly slow down the patient's heart rate below 50bpm for a few seconds. Therefore 6mg adenosine as a rapid i.v. bolus will be administered. The adenosine application will slow down the patient's heart rate and allow for correct mapping by the CIT device. Medical therapy of atrial fibrillation is started immediately according to local protocol. Since non-invasive mapping is performed within a few minutes, the therapy of atrial fibrillation will not be critically delayed. Consecutively, a low-dose thoracic computed tomography (CT) scan (neck to upper abdomen) will be performed independent from the patient's rhythm.
  Other Names: CardioInsightTM Cardiac Mapping System
Diagnostic Test: Computed tomography scan — The CT scans will follow a standardised protocol as predefined by the manufacturer of the CIT vest, Medtronic (Dublin, Ireland). After the sensor array has been placed on the patient, the patient is ready to undergo a CT scan to register each electrode's locations with respect to the body surface. All CT scans cover a body region from neck to the upper abdomen, have no cardiac gating performed or any contrast agent given. The CT scans are acquired on 3 CT scanners manufactured by Siemens Corporation (Berlin, Germany) with a fixed tube voltage of 80 kVp and 250 effective mAs (=mAs/pitch). The reconstruction parameters are of 3 mm slice thickness and of 1.5 mm increment (slice overlap) The estimated effective dose (ED) is 3.2 mSv per patient.

SUMMARY:
This study is to describe the exact location of NOAF-maintaining foci and rotors after cardiac surgery identified by mapping using the non-invasive phase mapping with CardioInsightTM - 3D Mapping technology (CardioInsightTM, Medtronic Switzerland, Tolochenaz, Switzerland) and a low-dose computed tomography scan of the chest.

DETAILED DESCRIPTION:
Atrial fibrillation (AF) is the most commonly oberserved postoperative complication after cardiac surgery. New-onset atrial fibrillation (NOAF) leads to prolonged intensive care unit (ICU) and hospital length of stay, increased early mortality and stroke along with higher treatment costs.

The exact location of structures triggering or maintaining NOAF is unknown. Identifying the exact location of NOAF- maintaining foci and rotors could allow development of preventive treatment strategies like preoperative ablation or perioperative ablation of high-risk foci. Non-invasive phase mapping with CardioInsightTM (CIT) - 3D Mapping technology (CardioInsightTM, Medtronic Switzerland, Tolochenaz, Switzerland) allows non-invasive description of AF foci and rotors with a 252-electrode vest applied to the patient's torso due to detailed mapping of NOAF-maintaining structures without invasive electrophysiological examination.

This study is to describe the exact location of NOAF-maintaining foci and rotors after cardiac surgery identified by mapping using the non-invasive phase mapping with CardioInsightTM - 3D Mapping technology (CardioInsightTM, Medtronic Switzerland, Tolochenaz, Switzerland) and a low-dose computed tomography scan of the chest.

ELIGIBILITY:
Inclusion Criteria:

* Cardiac surgery
* Signed informed consent by patient or next of kin

Mapping inclusion criteria

* NOAF within the first seven postoperative days (168 hours) after cardiac surgery developing on the cardiac surgery ward, intermediate care unit or the intensive care unit of the University Hospital Basel. ICU admission will be set as starting point for observation time.

General Exclusion Criteria:

Preoperative conditions:

* History of previous left atrial ablation
* History of cardioembolic stroke
* History of amiodarone treatment within three months
* Any documented history of atrial fibrillation/atrial flutter before surgery
* Left ventricular ejection fraction <40%
* Patient included into other study with radiation exposure

Perioperative conditions

* Perioperative mechanical circulatory support (e.g., intraaortic balloon pump; extracorporeal membrane oxygenation; left ventricular assist device (e.g. Impella, Abiomed Inc., Aachen, Germany)

Mapping exclusion criteria

* Heart rate ≥ 50 bpm AND contraindication to adenosine.

Contraindications to adenosine:

* Allergy/intolerance to adenosine
* History of chronic obstructive pulmonary disease (COPD Gold IV)(28)
* History of asthma
* History of Long-QT syndrome
* Hemodynamically unstable patients (margin of discretion of the attending physician)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Ongoing recruitment of elective and emergent patients through the study team will be performed during daily practice. All patients referred to the Department of Cardiac Surgery, University Hospital Basel, are routinely informed about the potential complication of NOAF. Besides, patients are informed about the BigMap study, mapping with CIT, its indications and contraindications. All patients who have given informed consent before surgery and present with NOAF are monitored and the mapping procedure is performed.
Sampling Method: Probability Sample
Enrollment: 157 (Estimated)
Dates: Start 2022-04-12 (Actual); Primary Completion 2028-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
localisation of foci and rotors maintaining NOAF after cardiac surgery identified by mapping | one time assessment at baseline (up to 5 minutes)
  localisation of foci and rotors maintaining NOAF after cardiac surgery identified by mapping system as three-dimensional electroanatomic map of the heart.

CONTACTS AND LOCATIONS:
Overall Officials: David Santer, Dr. med., Principal Investigator — Department of Cardiac Surgery, University Hospital Basel; Martin Siegemund, Prof. Dr. med., Study Director — Department of Cardiac Surgery, University Hospital Basel
Locations (2):
- University Hospital St. Pölten, Sankt Pölten, Austria
- Department of Cardiac Surgery, University Hospital Basel, Basel, Switzerland